CLINICAL TRIAL: NCT04983966
Title: Comparison of Quality of Recovery (QoR)-15 Scores According to the Anesthetics (Desflurane vs. Remimazolam) in the Patients With Lumbar Fusion Surgery: a Prospective Double-blind Randomized Controlled Trial
Brief Title: Comparison of Postoperative QoR-15 Scores Between Desflurane and Remimazolam in Lumbar Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Myoung Hwa Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3-2021-0214
Record Dates: First submitted 2021-07-28; First posted 2021-07-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Lumbar Fusion Surgery
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane group (Experimental): General anesthesia with volatile agent of desflurane
  Interventions: Drug: Desﬂurane
- Remimazolam group (Active Comparator): Remimazolam group will be started with remiamazolam at 6 mg/kg/h and TCI Minto model of remifentanil for the time of anesthesia induction, and maintained at 0.5-1.5 mg/kg/h.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Desﬂurane — General anesthesia for patients will be inducted and maintained with desflurane inhalation and remifentanil infusion.
  Remimazolam group will be started with remiamazolam at 6 mg/kg/h and TCI Minto model of remifentanil for the time of anesthesia induction, and maintained at 0.5
  Arms: Desflurane group
Drug: Remimazolam — General anesthesia for patients will be inducted and maintained with desflurane inhalation and remifentanil infusion.
  Remimazolam group will be started with remiamazolam at 6 mg/kg/h and TCI Minto model of remifentanil for the time of anesthesia induction, and maintained at 0.5
  Arms: Remimazolam group

SUMMARY:
The purpose of the study is to compare the quality of recovery (QoR)-15 scores according to the use of maintenance anesthetics in the lumbar fusion surgery. Total intravenous anesthesia (TIVA) have been known to help reducing risks of postoperative nausea/vomiting and malignant hyperthermia. However, it is still not enough to explain which is better between TIVA or inhalation anesthesia. In particular, there is no study to investigate overall postoperative functional recovery via QoR-15 in patients receiving TIVA with remimazolam. The hypothesis of our study is that total intravenous anesthesia based on remimazolam will demonstrate better quality of recovery compared with the anesthesia based on inhalation using desflurane.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients who aged 20-70 years with ASA-PS 1-3, BMI <30 undergoing lumbar fusion surgery under general anesthesia

Exclusion Criteria:

* Tolerance or hypersensitivity to benzodiazepine or propofol
* Dependence or addiction to psychotropic drugs or alcohol
* Pregnant women
* subjects who lack the ability to make decisions and susceptible to voluntary participation decisions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
The difference of QoR-15 scores | postoperative day 1
  The difference of scores in the Quality of Recovery (QoR)-15 survey between desflurane group and remimazolam group. 0 (minimum), 150 (maximum): Higher scores means better.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided